CLINICAL TRIAL: NCT00875043
Title: A Pilot Study to Determine the Effect on Intraocular Pressure, Optic Nerve Imaging and Other Markers of Venous Congestion of Volunteer Subjects in the Prone Position for a Period of Five Hours
Brief Title: Determine the Effect of Intraocular Pressure (IOP), Optic Nerve Imaging, Venous Congestion in Volunteers Prone Position 5 Hours
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Anesthesia Patient Safety Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 0120070324
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2009-04

CONDITIONS: Blindness
Keywords: ischemic optic neuropathy; cortical blindness
MeSH Terms: conditions — Blindness; Optic Neuropathy, Ischemic; Blindness, Cortical

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. flat Jackson table: All measurements previously described will be done with the patient in the prone postion and Jackson table flat.
- 2. Elevated Jackson tablet: All measurements previously described will be performed with subjects placed prone on the elevated Jackson table.

SUMMARY:
The purpose of this study is to provide data that would give the investigators a better understanding of the physiologic changes that occur and may contribute to post operative blindness. An improved understanding may lead to the development of protocols or devices that reduce the chance of catastrophic visual loss.

DETAILED DESCRIPTION:
Post operative vision loss resulting from nonocular surgery is a devastating, poorly understood and potentially preventable complication. Ischemic optic neuropathy, affecting both the anterior or posterioir portions of the optic nerve, is the most common cause of postoperative vision loss(POVL). Other, less common causes include retinal artery occlusion, retinal vein occlusion, retinal embolism, and cortical blindness. The estimated incidence of POVL in patients undergoing general anesthesia is 1/60,000. The incidence dramatically increases in cardiopulmonary bypass and prone spine surgery with estimates at 1/1600 and 1/1100, respectively. The etiology is unknown but it is thought to be multifactorial, and several potential risk factors have been identified, including degree of hypotension, preoperative hematocrit, external compression of the eye, blood loss and prone position. The investigators are proposing eight volunteers in two different sessions of 5.5 hours each. The first session the volunteer will lie prone of the flat Jackson table and the second session the volunteer will spend 5 hours prone on the Jackson table with a table elevation of 6 inches. The following measurements will be done: Intraocular Pressure (IOP) with a device called the Tonopen-XL, the Nidex NM 200 to visualize the retinal optic nerve imaging, refractometry, ultrasound, corneal thickness pachymetry, measurement of proptosis, measurement of pupillary reflex, The volunteers do not receive anesthetic medications or intravenous fluids and will provide a baseline for comparision with patients enrolled in the prospective study.

ELIGIBILITY:
Inclusion Criteria:

* subjects willing to consent

Exclusion Criteria:

* individuals unable to tolerate prone position for 5 hours
* individuals unable to tolerate contact lens placement
* females who are pregnant
* individuals with a sensitivity to proparacaine hcl 0.5% or tropicamide 1%
* individuals who are unable to have repeated mesaurements of intaocular pressure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geordie P. Grant, MD, Principal Investigator — University of Medicine & Dentistry of New Jersey
Locations (1):
- UMDNJ/University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No